CLINICAL TRIAL: NCT06413173
Title: Remotely Supervised tDCS Combined With Cognitive Training to Improve Complex Attention in Active Duty Service Members and Veterans With Mild TBI (Cognetric)
Brief Title: Remotely Supervised tDCS+ for Complex Attention in mTBI (Cognetric)
Acronym: COGNETRIC
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: United States Naval Medical Center, San Diego (U.S. Federal Agency)
Collaborators: Minneapolis Veterans Affairs Medical Center (U.S. Federal Agency); University of Minnesota (Other); United States Department of Defense (U.S. Federal Agency); Center for Veterans Research and Education (Other); The Defense and Veterans Brain Injury Center (U.S. Federal Agency); General Dynamics Information Technology (Unknown)
Responsible Party: Principal Investigator, Lars Hungerford, Senior Clinical Research Director, United States Naval Medical Center, San Diego
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: NMCSD.2023.0048
Record Dates: First submitted 2024-04-30; First posted 2024-05-14 (Actual); Last update posted 2025-11-12 (Actual); Status verified 2025-11

CONDITIONS: Brain Concussion; Brain Trauma; Attention Concentration Difficulty; Brain Injuries; Brain Injuries, Traumatic; Neurocognitive Dysfunction; Attention Impaired; Memory Impairment; Mild Traumatic Brain Injury; Mild Cognitive Impairment; Post Concussive Symptoms
Keywords: Military Health; Brain Stimulation; Cognitive Training; Cognitive Rehabilitation; Telehealth; Neuromodulation
MeSH Terms: conditions — Brain Concussion; Brain Injuries, Traumatic; Brain Injuries; Cognition Disorders; Memory Disorders; Cognitive Dysfunction; Post-Concussion Syndrome

STUDY DESIGN:
Intervention Model Description: This is a double-blind, randomized, placebo (sham) controlled pilot study.
Who Masked: Participant, Care Provider, Investigator
Masking Description: The tDCS unit software has a double-blind selection, blinding all study members, care providers, and participants until blinds are broken.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active tDCS (Experimental): Participants will receive 10 sessions of cognitive training concurrent with transcranial direct current stimulation. Stimulation will be applied for 20 minutes at the beginning of each session. Current will be ramped from 0 mA to 2 mA over 30 seconds, and then ramped down from 2 mA to 0 mA at the end of 20 minutes. Current will be applied via two electrodes consisting of a pre-inserted carbon rubber snap electrode that is pre-saturated with saline and connects directly to designated electrode sites located on the tDCS headband. The anodal stimulating electrode will be at location F3 (based on the 10-20 EEG location system) and the cathodal electrode at location F4.
  Interventions: Combination Product: Active tDCS and Cognitive Training Intervention
- Sham tDCS (Sham Comparator): Electrodes will be placed at the same positions as for active stimulation (F3 and F4), but current will be ramped down immediately after the initial 30s ramp up period and then at 20 minutes ramped up and down as done at the beginning. Thus, participants feel the initial tingling sensation associated with tDCS, but will receive no active current for the rest of the stimulation period
  Interventions: Combination Product: Sham tDCS and Cognitive Training Intervention

INTERVENTIONS:
Combination Product: Active tDCS and Cognitive Training Intervention — Cognitive training will occur concurrently with active tDCS session. The cognitive training occurs on a computer and consists of 5 exercises specifically selected and scientifically supported to (i) place demands on the executive function system (e.g. working memory, behavioral inhibition, decision making, and set- shifting), (ii) adapt to challenge the participant's current ability level, (iii) provide ongoing feedback, and (iv) present novel stimuli across visual and auditory modalities During each 45-minute training period, participants will complete the daily assigned adaptive training module. Following the completion of training sessions 1, 5, and 10, participants will be asked to supply a subjective workload assessment.
  Arms: Active tDCS
Combination Product: Sham tDCS and Cognitive Training Intervention — Cognitive training will occur concurrently with sham tDCS session. The cognitive training occurs on a computer and consists of 5 exercises specifically selected and scientifically supported to (i) place demands on the executive function system (e.g. working memory, behavioral inhibition, decision making, and set- shifting), (ii) adapt to challenge the participant's current ability level, (iii) provide ongoing feedback, and (iv) present novel stimuli across visual and auditory modalities During each 45-minute training period, participants will complete the daily assigned adaptive training module. Following the completion of training sessions 1, 5, and 10, participants will be asked to supply a subjective workload assessment.
  Arms: Sham tDCS

SUMMARY:
The proposed study will evaluate a new approach to cognitive rehabilitation of mTBI using a brain stimulation technique called "Remotely Supervised Transcranial Direct Current Stimulation combined with Cognitive Training" (RS-tDCS+) which has shown promise for improving complex attention in both healthy and clinical populations. RS-tDCS+ is a home-based, low-risk, non-invasive technique that is designed to boost cognitive training by enhancing learning and the brain's ability to reorganize connections. This study will evaluate RS-tDCS+ for improving complex attention in Active Duty Service Members (ADSM) and Veterans with a history of mTBI. Different tests of complex attention and symptom questionnaires will be used to determine the effects of real versus sham (placebo) RS-tDCS+. Second, the investigators will investigate electrical and connectivity changes in the brain associated with RS-tDCS+ using electroencephalogram (EEG) and magnetic resonance imaging (MRI). Third, the investigators will investigate the lasting effects of any observed changes by evaluating participants at 1 and 6 weeks post-treatment. Lastly, the investigators will explore the impact of individual differences (e.g., PTSD, depression, sleep quality, time since injury, baseline impairment, age, sex, ADSM versus Veteran) on treatment outcome.

DETAILED DESCRIPTION:
Objectives:

Attention, concentration, and working memory (i.e., complex attention) deficits are the most reported neurocognitive sequelae of mild traumatic brain injury (mTBI) and have been associated with patterns of decreased neural activation. Existing cognitive rehabilitation interventions require significant time and effort and are limited by small-to-moderate effect sizes and uncertain durability/generalization of effects. Novel, neuroplasticity-based interventions that improve complex attention and can be administered remotely are needed to increase access to care, decrease recovery time, and improve outcomes and quality of life following mTBI. This multi-site study will investigate remotely-supervised tDCS (RS-tDCS) combined with cognitive training in the chronic phase of recovery (≥3 months) from mTBI to 1) increase accessibility to care, 2) improve cognitive functioning, post-concussion symptom outcomes, and quality of life and 3) investigate the durability of the intervention in Active Duty Service Members (ADSM; at the Naval Medical Center San Diego (NMCSD) and Veterans (at the Minneapolis VA Health care System (MVAHCS)).

Research Plan and Methods:

This is a double-blind, randomized, sham-controlled study. 80 Veterans from the MVAHCS and 80 ADSM from NMCSD (total N=160) will be recruited. Participants will have a history of mTBI and self-reported attention and/or concentration difficulties. Baseline assessment will include self-reported symptoms and objective neurocognitive performance. Resting state functional connectivity changes will be measured with functional magnetic resonance imaging (fMRI) and oscillatory brain activity will be measured with EEG, both collected at baseline and at post-intervention assessments. Participants will be randomized to either active RS-tDCS or sham RS-tDCS, using stratified randomization by baseline cognitive scores. The intervention sessions will occur in the participant's home, 10 sessions within 2 weeks. Two post-intervention assessments, mirroring the baseline assessment, will occur approximately 1 week and 6 weeks after the intervention. Additionally, the investigators will collect longitudinal real-time data, daily, on TBI symptoms, cognitive, and mood factors during the 6 weeks post-intervention using Ecological Momentary Assessment (EMA).

Clinical Relevance:

RS-tDCS+ addresses two major obstacles of current TBI treatments: Accessibility and adherence. RS-tDCS+ offers several benefits as it can be monitored remotely, and can be self-administered in the home after the first session. If RS-tDCS proves effective, this non-invasive intervention could dramatically improve access to a validated treatment that can be rapidly implemented within various DOD and VA settings to reduce TBI-related symptoms, improve cognition, enhance recovery, bolster occupational performance, and improve quality of life.

ELIGIBILITY:
Inclusion Criteria:

1. Active-Duty Service Members.
2. Ages 18 to 60.
3. All genders.
4. All racial and ethnic groups.
5. History of mild TBI (as defined by the DOD/VA criteria used in conjunction with the OSU TBI-ID) sustained at least 3 months and no more than 10 years prior to enrollment.
6. Self-reported attention and/or concentration difficulties.
7. At least one cognitive symptom reported on the Neurobehavioral Symptom Inventory (NSI) cognitive subscale.

Exclusion Criteria:

1. Presence of a medical, psychiatric, physical or non-physical disease, disorder, condition, injury, disability or pre-existent history such that study participation, in the opinion of the PI: (a) may pose a significant risk to the participant; (b) raises the possibility that the participant is unlikely to successfully complete all of the requirements of the study according to the study protocol; or (c) might adversely impact the integrity of the data or the validity of the study results. Specific conditions include (but are not limited to) a history of: brain tumor, epilepsy, cerebral vascular accident (CVA), Schizophrenia, Bipolar Disorder, and Mania.
2. History of prior treatment with ECT or neuromodulation in the last 12 months.
3. Current, diagnosed substance dependence.
4. Newly prescribed medication within the previous 3 weeks.
5. Diagnosis of intellectual disability or pervasive developmental disorder (i.e., premorbid IQ less than or equal to 70).
6. Any medical condition or treatment other than mild TBI (e.g., stroke, tumor, HIV, moderate-severe TBI), with significant neurological disorder or insults that, based on the Principal Investigator's judgment, would impact risk.
7. Psychosis or mania within 30 days of enrollment, as determined by the PI, based on a psychiatric history and examination and/or a review of available medical records
8. Contraindications for tDCS (e.g., metallic cranial plates/screws or implanted device, eczema or skin lesions on scalp)
9. A positive pregnancy report.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 160 (Estimated)
Dates: Start 2024-07-25 (Actual); Primary Completion 2028-09-30 (Estimated); Study Completion 2028-09-30 (Estimated)

PRIMARY OUTCOMES:
Symbol Digit Modalities Test (SDMT) | Baseline, 1-week post, & 6-weeks post intervention
  Standardized neuropsychological assessment measure of visual attention and working memory
Neuropsychological Assessment Battery (NAB) Attention Module | Baseline, 1-week post, & 6-weeks post intervention
  Standardized neuropsychological assessment consisting of 4 subtests to assess visual and auditory attention, working memory, and scanning
Neurobehavioral Symptom Inventory (NSI) | Baseline, 1-week post, & 6-weeks post intervention
  A measure of common post-concussive symptoms rated on a 5-point Likert scale (0-4); with low scores corresponding to mild or no incidence of symptoms and high scores corresponding to more severe incidence of symptoms.
Electroencephalogram (EEG) - Resting State Functional Connectivity | Baseline, 1-week post, & 6-weeks post intervention
  Resting State EEG will be collected to assess neural dynamics or functional connectivity and spectral power of delta,theta, alpha, beta, and gamma frequency bands.
Electroencephalogram (EEG) - Resting State Spectral Power | Baseline, 1-week post, & 6-weeks post intervention
  Resting State EEG will be collected to assess spectral power of standard frequency bands (delta, theta, alpha, beta, and gamma).
Magnetic Resonance Imaging (MRI) - T1 (optional) | Baseline & 1-week post intervention
  MRI will be used to collect a T1-weighted (structural scan) pulse sequence of the brain.
Magnetic Resonance Imaging (MRI) - T2 (optional) | Baseline & 1-week post intervention
  MRI will be used to collect a T2-weighted pulse sequence of the brain.
Magnetic Resonance Imaging (MRI) - T2* (optional) | Baseline & 1-week post intervention
  MRI will be used to collect a T2*-weighted (BOLD-contrast fMRI / Resting State) pulse sequence of the brain.
Magnetic Resonance Imaging (MRI) - DWI (optional) | Baseline & 1-week post intervention
  MRI will be used to collect a Diffusion Weighted Imaging (DWI) pulse sequence of the brain (white-matter tractography).
Magnetic Resonance Imaging (MRI) - ASL (optional) | Baseline & 1-week post intervention
  MRI will be used to collect an Arterial Spin Labeling (ASL / Blood Flow Rate) pulse sequence of the brain.
Magnetic Resonance Imaging (MRI) - ROI Analysis (optional) | Baseline & 1-week post intervention
  T2*-weighted (Resting State) images will be analyzed with Region of Interest (ROI) time-courses to generate a partial correlation value (Fisher Z) that depicts functional connectivity.
NIH Toolbox Quality of Life Assessment (NeuroQoL) | Baseline, 1-week post, & 6-weeks post intervention
  Questionnaire to assess quality of life with regard to cognitive, social, emotional, and behavioral abilities rated on a 5-point Likert scale (1-5); with low scores corresponding to mild to no impairment in these abilities and high scores corresponding to more severe impairment in these abilities.
Insomnia Severity Index (ISI) | Baseline, 1-week post, & 6-weeks post intervention
  Measure of insomnia severity rated on a 5-point Likert scale (0-4); with low scores corresponding to mild or no incidence of insomnia and high scores corresponding to more severe incidences of insomnia.
Patient Health Questionnaire (PHQ-8) | Baseline, 1-week post, & 6-weeks post intervention
  The PHQ is a self-report inventory that is used as a screening and diagnostic tool for depressive disorders using a 4-point Likert scale (e.g., 0 = not at all, 3 = nearly every day), yielding a total score from 0 - 21. The eight-item Patient Health Questionnaire depression scale (PHQ-8) is established as a valid diagnostic and severity measure for depressive disorders in large clinical research studies.
PTSD Checklist- Civilian Version (PCL-C) | Baseline, 1-week post, & 6-weeks post intervention
  A 17-item self-report rating scale used as a screening tool for posttraumatic stress disorder (PTSD) using a 5-point Likert scale (e.g., 1 = not at all, 5 = extremely), yielding a total score from 17 - 85. This version asks about symptoms in relation to generic "stressful experiences" and can be used with any population. It simplifies assessment based on multiple traumas because symptom endorsements are not attributed to a specific event. Importantly, the PCL-C has been established as a valid measure of PTSD severity in Active Duty Service Members and Veterans.
Patient Global Impression of Change (PGIC) | 1-week post & 6-weeks post intervention
  This scale evaluates all aspects of patients' health and assesses if there has been an improvement or decline in clinical status. Specifically, individuals are asked to calculate the difference between their current and previous health state based on a Likert scale. They are required to answer the question "Since beginning treatment at this clinic, how would you describe the change (if any) in activity limitations, symptoms, emotions, and overall quality of life, related to your painful condition." Score ranges from 1 (no change or condition got worse) to 7 (a great deal better). They are then required to circle a number between 0 to 10 that reflects the degree of change since the start of the intervention. The test takes approximately 2 minutes to complete.
Information Sampling Task (IST) | Baseline, 1-week post, & 6-weeks post intervention
  A test of reflection impulsivity. It presents a series of trials with an array of 25 grey boxes arranged in a 5x5 matrix. The grey boxes conceal yellow or blue squares on each trial. The subject decides which of the two underlying colors (yellow or blue) lay in the majority. The subject can open as many boxes as they wish to make a decision. Correct decisions are awarded a number of points.
Groton Maze Learning Task (GMLT) | Baseline, 1-week post, & 6-weeks post intervention
  A cognitive test of spatial working memory and error monitoring that has been shown to be sensitive to detecting longitudinal change in cognitive ability.78 It consists of a 10 x 10 grid of grey tiles. To complete the maze, the participant must click on the tiles to follow a hidden pathway through the grid from the top left corner to the bottom right corner. They must only click on adjacent tiles, and return to the previous tile if an error is made before moving on. The participant receives visual and auditory feedback for correct and incorrect moves. There are various types of errors (e.g., perseverative error, rule-break error) recorded depending on which type of rule has been broken, and the time to complete the maze is recorded. The trial ends once the participant reaches the bottom right corner of the grid of tiles.
Fusion Task: BEAM | Baseline, 1-week post, & 6-weeks post intervention
  For the BEAM subtask, the subject will be directed to change his/her fixation from a crosshair displayed at the center of screen to a white circle appearing randomly on the left or right side of the screen. The subject will press a button labeled either "Left" or "Right" based on whether the circle appeared on the left or right of the screen. In a small percentage of the trials in which a red arrow appears in the center of the screen, the subject will be instructed not to look at the circle nor press any buttons (inhibition test). Saccadic eye movements, pupil responses, and manual response time (RT) in addition to errors will be recorded.
Fusion Task: N-Back | Baseline, 1-week post, & 6-weeks post intervention
  For the N-Back subtask, the subject will be directed to change his/her fixation from a cross sign displayed at the center of screen to a colored circle (Green or Blue) that randomly appears on the left or right side of the screen. In the first, '0-back' condition, the subject shall push a response button labeled either (1) "GREEN" or (2) "BLUE" in accordance with the color of the circle currently on the screen. In the second, '1-back' condition, immediately upon recognition of the color of the circle, the subject shall push a response button labeled with either (1) "SAME" if the color matches the circle that appeared previously, or (2) "DIFFERENT" if the color does not match. Saccadic eye movements, pupil responses, and manual response time (RT) in addition to errors will be recorded.
tDCS Symptom Rating Questionnaire (SRQ) | Assessment collected daily during the intervention block (b/t baseline & 1-week post)
  Questionnaire to assess pre-post tDCS symptom rating, rated on a 4-point Likert scale (0-3); with low scores corresponding to mild or no incidence of symptoms and high scores corresponding to severe incidence of symptoms.
Ecological Momentary Assessment (EMA) | Assessment collected daily during the intervention block (b/t baseline & 1-week post)
  A data capture technique that involves repeated sampling of thoughts, feelings, or behaviors as close in time to the experience as possible in the naturalistic environment. A series of 18 self-report questions rated on a 10-point Likert scale (Q1 - Q15) and 5-point Likert scale (Q16 - Q18) regarding mood, current cognitive state, and environment. EMA data is used to look for relationships between variables with the causal discovery analysis.

SECONDARY OUTCOMES:
BrainHQ Task Load Index (TLX) | Collected during the Intervention block at sessions 1, 5, & 10 (b/t baseline & 1-week post)
  Subjective workload assessment of level of effort, mental demand, frustration, and performance during cognitive training, rated on a 10-point Likert scale (1-10); with low scores corresponding to less effort or mental demand and high scores corresponding to more effort or mental demand.
Fusion Task Load Index (F-TLX) | Baseline, 1-week post, & 6-weeks post intervention
  An assessment tool that rates perceived workload to assess a participant's ability and level of performance on the sub-components of the Fusion task. Participants will answer questions regarding their level of effort, mental demand, frustration, physical demand, temporal demand, and performance on each task.

CONTACTS AND LOCATIONS:
Overall Officials: Lars D Hungerford, PhD, Principal Investigator — United States Naval Medical Center, San Diego
Locations (2):
- United States (2):
  - Naval Medical Center San Diego, San Diego, California
  - Minneapolis VA Health Case System, Minneapolis, Minnesota

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Informed Consent Form (2023-11-01): https://cdn.clinicaltrials.gov/large-docs/73/NCT06413173/ICF_000.pdf